CLINICAL TRIAL: NCT05318820
Title: A Phase I Monocentric, Open-label, Randomized, Crossover Clinical Study to Evaluate the Pharmacokinetics and Bioequivalence of HMPL-523 Tablets Produced by Two Different Manufacturers in Healthy Chinese Subjects
Brief Title: A Clinical Study to Evaluate the Pharmacokinetics and Bioequivalence of HMPL-523 Tablets Produced by Two Different Manufacturers
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Hutchison Medipharma Limited (Industry)
Responsible Party: Sponsor
Organization: Hutchmed (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2021-523-00CH1
Record Dates: First submitted 2022-03-09; First posted 2022-04-08 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Healthy Subject

STUDY DESIGN:
Intervention Model Description: This is a monocentric, randomized, open-label, single-dose, three-cycle, partial replicate clinical study designed to evaluate the pharmacokinetic profile and bioequivalence of HMPL-523 Tablets produced by two different manufacturers in healthy subjects. This study plans to enroll 39 healthy Chinese subjects who will be randomized (1:1:1) into one of three sequence groups (Test [T]/Reference[R]/R group, RTR group and RRT group) to receive a single dose in each cycle with a washout period of at least 7 days, where T is the test product [i.e., HMPL-523 Tablets manufactured by Hutchison MediPharma (Suzhou) Limited.], and R is the reference product (i.e., HMPL-523 Tablets manufactured by WuXi STA).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HMPL-523-TRR (Experimental): Three cycle dose: TRR Test product: HMPL-523 Tablets manufactured by Hutchison MediPharma (Suzhou) Co., Ltd.; Reference product: HMPL-523 Tablets manufactured by WuXi STA
  Interventions: Drug: HMPL-523
- HMPL-523-RTR (Experimental): Three cycle dose:RTR Test product: HMPL-523 Tablets manufactured by Hutchison MediPharma (Suzhou) Co., Ltd.; Reference product: HMPL-523 Tablets manufactured by WuXi STA
  Interventions: Drug: HMPL-523
- HMPL-523-RRT (Experimental): Three cycle dose:RRT Test product: HMPL-523 Tablets manufactured by Hutchison MediPharma (Suzhou) Co., Ltd.; Reference product: HMPL-523 Tablets manufactured by WuXi STA
  Interventions: Drug: HMPL-523

INTERVENTIONS:
Drug: HMPL-523 — This study plans to enroll 39 healthy Chinese subjects who will be randomized (1:1:1) into one of three sequence groups (Test [T]/Reference[R]/R group, RTR group and RRT group) to receive a single dose in each cycle with a washout period of at least 7 days, where T is the test product [i.e., HMPL-523 Tablets manufactured by Hutchison MediPharma (Suzhou) Limited.], and R is the reference product (i.e., HMPL-523 Tablets manufactured by WuXi STA).

SUMMARY:
This is a monocentric, randomized, open-label, single-dose, three-cycle, partial replicate clinical study designed to evaluate the pharmacokinetic profile and bioequivalence of HMPL-523 Tablets produced by two different manufacturers in healthy subjects.

DETAILED DESCRIPTION:
This is a monocentric, randomized, open-label, single-dose, three-cycle, partial replicate clinical study designed to evaluate the pharmacokinetic profile and bioequivalence of HMPL-523 Tablets produced by two different manufacturers in healthy subjects. This study plans to enroll 39 healthy Chinese subjects who will be randomized (1:1:1) into one of three sequence groups (Test [T]/Reference[R]/R group, RTR group and RRT group) to receive a single dose in each cycle with a washout period of at least 7 days, where T is the test product [i.e., HMPL-523 Tablets manufactured by Hutchison MediPharma (Suzhou) Limited.], and R is the reference product (i.e., HMPL-523 Tablets manufactured by WuXi STA).

The study includes three periods expected to last for 2 months: screening period, treatment period (for three cycles), and follow-up period

ELIGIBILITY:
Inclusion Criteria:

1. Subjects can communicate well with investigators, must be voluntary and sign the ICF, and agree to comply with the requirements in the study protocol;
2. Healthy male and female subjects aged 18-55 years (inclusive);
3. Weight ≥50 kg, Body Mass Index (BMI) between 19-26 kg/m2 (inclusive);
4. Subjects with good health condition
5. Subjects of childbearing potential must promise to use reliable contraceptive measures.

Exclusion Criteria:

1. History or clinical characterization of clinically significant metabolic/endocrine, hepatic, renal, hematological, pulmonary, immune, cardiovascular, gastrointestinal, genitourinary, neurological, or psychiatric diseases within 3 months prior to the screening period and in the screening period (judged by investigators);
2. creatinine clearance estimated using Cockcroft-Gault formula [(140-age) × body weight (kg) × gender correction factor] /[0.818×Scr (umol/L)] (male: 1.00, female: 0.85) < 80 mL/min;
3. History of gastrointestinal surgery, kidney surgery, cholecystectomy and other surgeries that might affect drug absorption or excretion judged by the investigator;
4. History of serious allergy (e.g., drug allergy) and acute allergic rhinitis or food allergy, in particular allergy to the active ingredient or excipient of study drug, within two weeks prior to screening;
5. Previous history of hypertension;
6. Systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg;
7. Female subjects who have a positive pregnancy test;
8. Subjects who smoked >10 cigarettes per day within 3 months prior to screening, or are unable to quit smoking completely during the study;
9. Subjects who drank on a regular basis within 6 months prior to the study, i.e., drinking more than 14 units of alcohol per week (1 unit =360 mL beer or 45 mL liquor with 40% alcohol or 150 mL wine);
10. Subjects with drug abuse (including but not limited to Morphine, 3,4-methylenedioxy-methamphetamine (MDMA), methamphetamine, tetrahydrocannabinolic acid, Ketamine, Cocaine or subjects whose urine drug abuse screen showed positive);
11. Use of blood products within 2 months before screening; donation of blood (including blood component) or loss of blood ≥400 mL within 3 months prior to screening, ≥200 mL within 1 month prior to screening, or plan to donate blood or blood component during the study or within 1 month after end of the study;
12. Subjects who have a fear of needles, hemophobia or whose venous blood is hard to collect;
13. Positive test for hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb), hepatitis C virus (HCV) antibody, human immunodeficiency virus (HIV) antibody, or treponema pallidum antibody;
14. Use of any prescription drug and Chinese herbal tonic within 30 days prior to the first dose;
15. Use of any over-the-counter drug (including but not limited to vitamins, prophylactic treatments, plant health products, etc.) within 14 days prior to the first dose;
16. Having participated in clinical trials for other drugs/medical devices within 3 months prior to screening;
17. Having consumed foods, juices and beverages containing alcohol, grapefruit, bigarade and caffeine within 72 hours prior to the first dose;
18. Subjects vaccinated with a live-attenuated vaccine within 8 weeks prior to screening or planning to get vaccinated during participation of this clinical trial;
19. Previous history of serious gastrointestinal disease, such as dysphagia, active gastric ulcer, inability to take drugs orally or absorption disorder for oral drugs;
20. Subjects who have special requirements for diet and cannot comply with uniform diet;
21. Lactating female subjects;
22. According to the investigator's judgment, the subjects had any other disease or status that might affect the normal completion of the study or the evaluation of the study data, or had any other condition that was not suitable for the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
maximum plasma concentration (Cmax) | through study completion, an average of 2 months
  To evaluate the pharmacokinetics and bioequivalence of HMPL- 523 Tablets 300 mg (100 mg/tablet×3) (produced by two different manufacturers) taken orally in a single dose after a standard meal in healthy Chinese subjects
time to maximum plasma concentration (Tmax) | Time Frame: through study completion, an average of 2 months
  To evaluate the pharmacokinetics and bioequivalence of HMPL- 523 Tablets 300 mg (100 mg/tablet×3) (produced by two different manufacturers) taken orally in a single dose after a standard meal in healthy Chinese subjects
terminal elimination half-life (t1/2) | through study completion, an average of 2 months
  To evaluate the pharmacokinetics and bioequivalence of HMPL- 523 Tablets 300 mg (100 mg/tablet×3) (produced by two different manufacturers) taken orally in a single dose after a standard meal in healthy Chinese subjects
Area under plasma drug concentration-time curve (AUC0-t, AUC0-∞) | through study completion, an average of 2 months
  To evaluate the pharmacokinetics and bioequivalence of HMPL- 523 Tablets 300 mg (100 mg/tablet×3) (produced by two different manufacturers) taken orally in a single dose after a standard meal in healthy Chinese subjects

SECONDARY OUTCOMES:
Ratio between AUCs of two HMPL-523 Tablets | through study completion, an average of 2 months
  To compare the relative bioavailability of HMPL-523 Tablet 300 mg (100 mg/tablet ×3) produced by two different manufacturers
safety information/AE,SAE | through study completion, an average of 2 months
  To observe the safety of HMPL-523 Tablet 300 mg (100 mg/tablet ×3) taken orally in a single dose after a standard meal in healthy Chinese subjects

CONTACTS AND LOCATIONS:
Overall Officials: Jingying Jia, Principal Investigator — Shanghai Xuhui Central Hospital
Locations (1):
- Shanghai Xuhui Central Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No